CLINICAL TRIAL: NCT03759379
Title: HELIOS-A: A Phase 3 Global, Randomized, Open-label Study to Evaluate the Efficacy and Safety of ALN-TTRSC02 in Patients With Hereditary Transthyretin Amyloidosis (hATTR Amyloidosis)
Brief Title: HELIOS-A: A Study of Vutrisiran (ALN-TTRSC02) in Patients With Hereditary Transthyretin Amyloidosis (hATTR Amyloidosis)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALN-TTRSC02-002; 2023-508365-33-00 (EU CTIS Number); 2018-002098-23 (EudraCT Number)
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Results first posted 2022-08-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Amyloidosis, Hereditary; Transthyretin Amyloidosis
MeSH Terms: conditions — Amyloidosis, Familial; Amyloidosis, Hereditary, Transthyretin-Related | interventions — patisiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vutrisiran + Vutrisiran (HELIOS-A) (Experimental): Participants will receive vutrisiran 25 mg subcutaneous (SC) injection once every 3 months (q3M) for 18 months during the Treatment Period followed by vutrisiran 50 mg SC injection once every 6 months (q6M) or vutrisiran 25 mg q3M during the Randomized Treatment Extension (RTE) Period. Upon implementation of Amendment 6, participants receiving vutrisiran SC 50 mg q6M will transition to vutrisiran SC 25 mg q3M at their next scheduled dosing.
  Interventions: Drug: Vutrisiran
- Patisiran + Vutrisiran (HELIOS-A) (Active Comparator): Participants will receive patisiran 0.3 mg/kg intravenous (IV) infusion once every 3 weeks (q3w) for 18 months during the Treatment Period followed by vutrisiran 50 mg SC injection once q6M or vutrisiran 25 mg q3M during the RTE Period. Upon implementation of Amendment 6, participants receiving vutrisiran SC 50 mg q6M will transition to vutrisiran SC 25 mg q3M at their next scheduled dosing.
  Interventions: Drug: Patisiran; Drug: Vutrisiran

INTERVENTIONS:
Drug: Patisiran — Patisiran will be administered by IV infusion.
  Other Names: ONPATTRO; ALN-TTR02
  Arms: Patisiran + Vutrisiran (HELIOS-A)
Drug: Vutrisiran — Vutrisiran will be administered by SC injection.
  Other Names: ALN-TTRSC02; AMVUTTRA

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of vutrisiran (ALN-TTRSC02) in participants with hereditary transthyretin amyloidosis (hATTR amyloidosis). Participants will receive vutrisiran subcutaneous (SC) injection once every 3 months (q3M) or the reference comparator patisiran intravenous (IV) injection once every 3 weeks (q3w) during the 18 month Treatment Period. This study will use the placebo arm of the APOLLO study (NCT01960348) as an external comparator for the primary and most other efficacy endpoints during the 18 Month Treatment Period. Following the 18 Month Treatment Period, all participants will be randomized to receive vutrisiran 50 mg SC injection once every 6 months (q6M) or vutrisiran 25 mg q3M in the Randomized Treatment Extension (RTE) Period. Upon implementation of Amendment 6, participants receiving vutrisiran SC 50 mg q6M will transition to vutrisiran SC 25 mg q3M at their next scheduled dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of 18 to 85 years of age (inclusive);
* Has a diagnosis of hATTR amyloidosis with transthyretin (TTR) mutation;
* Has adequate neurologic impairment score (NIS);
* Has adequate polyneuropathy disability (PND) score;
* Has adequate Karnofsky Performance Status (KPS).

Exclusion Criteria:

* Had a prior liver transplant or is likely to undergo liver transplantation during the study;
* Has known other (non-hATTR) forms of amyloidosis or leptomeningeal amyloidosis;
* Has New York Heart Association heart failure classification >2;
* Clinically significant liver function test abnormalities;
* Has known human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV) infection;
* Received an experimental drug within 30 days of dosing;
* Received prior TTR-lowering treatment;
* Has other known causes of neuropathy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2025-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (61):
- United States (15):
  - Clinical Trial Site, La Mesa, California
  - Clinical Trial Site, Aurora, Colorado
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Fairway, Kansas
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Chapel Hill, North Carolina
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Portland, Oregon
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Dallas, Texas
- Clinical Trial Site, Buenos Aires, Argentina
- Australia (3):
  - Clinical Trial Site, Northmead, New South Wales
  - Clinical Trial Site, Brisbane, Queensland
  - Clinical Trial Site, Melbourne, Victoria
- Belgium (2):
  - Clinical Trial Site, Brussels
  - Clinical Trial Site, Leuven
- Clinical Trial Site, Rio de Janeiro, Brazil
- Clinical Trial Site, Sofia, Bulgaria
- Canada (2):
  - Clinical Trial Site, Montreal
  - Clinical Trial Site, Vancouver
- Clinical Trial Site, Nicosia, Cyprus
- France (6):
  - Clinical Trial Site, Bordeaux
  - Clinical Trial Site, Créteil
  - Clinical Trial Site, Le Kremlin-Bicêtre
  - Clinical Trial Site, Lille
  - Clinical Trial Site, Marseille
  - Clinical Trial Site, Nantes
- Germany (3):
  - Clinical Trial Site, Heidelberg
  - Clinical Trial Site, Mainz
  - Clinical Trial Site, Münster
- Clinical Trial Site, Athens, Greece
- Italy (4):
  - Clinical Trial Site, Messina
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Pavia
  - Clinical Trial Site, Rome
- Japan (4):
  - Clinical Trial Site, Kumamoto
  - Clinical Trial Site, Nagano
  - Clinical Trial Site, Nagoya
  - Clinical Trial Site, Osaka
- Clinical Trial Site, Kuala Lumpur, Malaysia
- Clinical Trial Site, Mexico City, Mexico City, Mexico
- Clinical Trial Site, Groningen, Netherlands
- Portugal (2):
  - Clinical Trial Site, Lisbon
  - Clinical Trial Site, Porto
- South Korea (2):
  - Clinical Trial Site, Daegu
  - Clinical Trial Site, Seoul
- Spain (5):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Hospitalet de Llobregat (Barcelona)
  - Clinical Trial Site, Huelva
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, Valencia
- Sweden (2):
  - Clinical Trial Site, Solna
  - Clinical Trial Site, Umeå
- Taiwan (2):
  - Clinical Trial Site, Taipei
  - Clinical Trial Site, Taoyuan
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Access to data may be declined where there is likelihood a patient could be identified or other feasibility issue, where there is a potential conflict of interest, a planned business activities or an actual or potential competitive risk. Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Timeframes for data access may vary and can take up to 6 months or more.
  Requests for access to data can be submitted via the website www.vivli.org. Questions can also be directed to datasharing@alnylam.com.

REFERENCES:
- [Derived] Luigetti M, Quan D, Berk JL, Conceicao I, Misumi Y, Chao CC, Bender S, Aldinc E, Vest J, Adams D. Impact of Baseline Neuropathy Severity on Vutrisiran Treatment Response in the Phase 3 HELIOS-A Study. Neurol Ther. 2024 Jun;13(3):625-639. doi: 10.1007/s40120-024-00595-9. Epub 2024 Mar 21. PMID 38512694
- [Derived] Obici L, Ajroud-Driss S, Lin KP, Berk JL, Gillmore JD, Kale P, Koike H, Danese D, Aldinc E, Chen C, Vest J, Adams D; HELIOS-A Collaborators Study Group. Impact of Vutrisiran on Quality of Life and Physical Function in Patients with Hereditary Transthyretin-Mediated Amyloidosis with Polyneuropathy. Neurol Ther. 2023 Oct;12(5):1759-1775. doi: 10.1007/s40120-023-00522-4. Epub 2023 Jul 31. PMID 37523143
- [Derived] Adams D, Tournev IL, Taylor MS, Coelho T, Plante-Bordeneuve V, Berk JL, Gonzalez-Duarte A, Gillmore JD, Low SC, Sekijima Y, Obici L, Chen C, Badri P, Arum SM, Vest J, Polydefkis M; HELIOS-A Collaborators. Efficacy and safety of vutrisiran for patients with hereditary transthyretin-mediated amyloidosis with polyneuropathy: a randomized clinical trial. Amyloid. 2023 Mar;30(1):1-9. doi: 10.1080/13506129.2022.2091985. Epub 2022 Jul 23. PMID 35875890

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with hATTR amyloidosis were enrolled and treated at 57 sites in Argentina, Australia, Belgium, Brazil, Bulgaria, Canada, Cyprus, France, Germany, Greece, Italy, Japan, Korea, Malaysia, Mexico, Netherlands, Portugal, Spain, Sweden, Taiwan, United Kingdom and United States. Data is reported for the 9-Month primary analysis period.
Pre-assignment Details: This study will use the placebo arm of the APOLLO study (NCT01960348) as an external comparator for the primary and most other efficacy endpoints (N=77).
Groups:
- Vutrisiran + Vutrisiran (HELIOS-A): Participants will receive vutrisiran 25 mg subcutaneous (SC) injection once every 3 months (q3M) for 18 months during the Treatment Period followed by vutrisiran SC injection once every 6 months (q6M) or q3M during the Randomized Treatment Extension (RTE) Period.
- Patisiran + Vutrisiran (HELIOS-A): Participants will receive patisiran 0.3 mg/kg intravenous (IV) infusion once every 3 weeks (q3w) for 18 months during the Treatment Period followed by vutrisiran SC injection q6M or q3M during the RTE Period.
Period: Treatment Period
Arm/Group | Vutrisiran + Vutrisiran (HELIOS-A) | Patisiran + Vutrisiran (HELIOS-A)
Started | 122 | 42
Completed | 0 | 0
Not Completed | 122 | 42
Not completed — Remained in this Period at Time of Data Cut | 119 | 38
Not completed — Death | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Period: Randomized Treatment Extension Period
Arm/Group | Vutrisiran + Vutrisiran (HELIOS-A) | Patisiran + Vutrisiran (HELIOS-A)
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who received any amount of study drug. Data from the placebo arm of the APOLLO study (NCT01960348) is included as it will be used as an external comparator for the primary and most other efficacy endpoints. The placebo APOLLO arm did not participate in this study.
Groups:
- External Placebo Comparator (APOLLO): Participants in the APOLLO study (NCT01960348) who received at least 1 dose of placebo.
- Vutrisiran + Vutrisiran (HELIOS-A): Participants will receive vutrisiran 25 mg SC injection q3M for 18 months during the Treatment Period followed by vutrisiran SC injection q6M or q3M during the RTE Period.
- Patisiran + Vutrisiran (HELIOS-A): Participants will receive patisiran 0.3 mg/kg IV infusion q3w for 18 months during the Treatment Period followed by vutrisiran SC injection q6M or q3M during the RTE Period.
- Total: Total of all reporting groups
Arm/Group | External Placebo Comparator (APOLLO) | Vutrisiran + Vutrisiran (HELIOS-A) | Patisiran + Vutrisiran (HELIOS-A) | Total
Number analyzed (Participants) | 77 | 122 | 42 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline characteristics data from the external placebo arm of the APOLLO study was not summarized with the data from HELIOS-A. APOLLO placebo data was only used as an external comparator for the primary and most other efficacy endpoints. Therefore APOLLO placebo baseline characteristic data is reported separately directly below.
  years
    number analyzed (Participants) | 0 | 122 | 42 | 164
    (all) |  | 57.8 (13.2) | 58.0 (10.5) | 57.9 (12.5)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline characteristics data from the external placebo arm of the APOLLO study was not summarized with the data from HELIOS-A. APOLLO placebo data was only used as an external comparator for the primary and most other efficacy endpoints. Therefore APOLLO placebo baseline characteristic data is reported separately.
  years
    number analyzed (Participants) | 77 | 0 | 0 | 77
    (all) | 62.2 (10.76) |  |  | 62.2 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics data from the external placebo arm of the APOLLO study was not summarized with the data from HELIOS-A. APOLLO placebo data was only used as an external comparator for the primary and most other efficacy endpoints. Therefore APOLLO placebo baseline characteristic data is reported separately directly below.
  Participants
    number analyzed (Participants) | 0 | 122 | 42 | 164
    Female |  | 43 | 15 | 58
    Male |  | 79 | 27 | 106
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics data from the external placebo arm of the APOLLO study was not summarized with the data from HELIOS-A. APOLLO placebo data was only used as an external comparator for the primary and most other efficacy endpoints. Therefore APOLLO placebo baseline characteristic data is reported separately.
  Participants
    number analyzed (Participants) | 77 | 0 | 0 | 77
    Female | 19 |  |  | 19
    Male | 58 |  |  | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics data from the external placebo arm of the APOLLO study was not summarized with the data from HELIOS-A. APOLLO placebo data was only used as an external comparator for the primary and most other efficacy endpoints. Therefore APOLLO placebo baseline characteristic data is reported separately directly below.
  Participants
    Asian: number analyzed (Participants) | 0 | 122 | 42 | 164
    Asian | 0 | 21 | 8 | 29
    Black or African American: number analyzed (Participants) | 0 | 122 | 42 | 164
    Black or African American | 0 | 4 | 4 | 8
    Multiple: number analyzed (Participants) | 0 | 122 | 42 | 164
    Multiple | 0 | 1 | 0 | 1
    Other: number analyzed (Participants) | 0 | 122 | 42 | 164
    Other | 0 | 10 | 1 | 11
    Unknown: number analyzed (Participants) | 0 | 122 | 42 | 164
    Unknown | 0 | 0 | 0 | 0
    White: number analyzed (Participants) | 0 | 122 | 42 | 164
    White | 0 | 86 | 29 | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics data from the external placebo arm of the APOLLO study was not summarized with the data from HELIOS-A. APOLLO placebo data was only used as an external comparator for the primary and most other efficacy endpoints. Therefore APOLLO placebo baseline characteristic data is reported separately.
  Participants
    Asian: number analyzed (Participants) | 77 | 0 | 0 | 77
    Asian | 25 |  |  | 25
    Black or African American: number analyzed (Participants) | 77 | 0 | 0 | 77
    Black or African American | 1 |  |  | 1
    White: number analyzed (Participants) | 77 | 0 | 0 | 77
    White | 50 |  |  | 50
    Unknown or Not Reported: number analyzed (Participants) | 77 | 0 | 0 | 77
    Unknown or Not Reported | 1 |  |  | 1
Modified Neuropathy Impairment Score +7 (mNIS+7) [Mean (Standard Deviation); unit: score on a scale] — The mNIS+7 is a composite score that measures neurologic impairment which includes the following components: physical exam of lower limbs, upper limbs and cranial nerves to assess motor strength/weakness, electrophysiologic measurement of small and large nerve fiber function, sensory testing and postural blood pressure. The mNIS+7 is scored from 0 (no impairment) to 304 points (maximum impairment). A higher score indicates a worse outcome. Population: Baseline characteristics data from the external placebo arm of the APOLLO study was not summarized with the data from HELIOS-A. APOLLO placebo data was only used as an external comparator for the primary and most other efficacy endpoints. Therefore APOLLO placebo baseline characteristic data is reported separately directly below.
  score on a scale
    number analyzed (Participants) | 0 | 122 | 42 | 164
    (all) |  | 60.55 (35.99) | 57.69 (33.71) | 59.82 (35.34)
Modified Neuropathy Impairment Score +7 (mNIS+7) [Mean (Standard Deviation); unit: score on a scale] — The mNIS+7 is a composite score that measures neurologic impairment which includes the following components: physical exam of lower limbs, upper limbs and cranial nerves to assess motor strength/weakness, electrophysiologic measurement of small and large nerve fiber function, sensory testing and postural blood pressure. The mNIS+7 is scored from 0 (no impairment) to 304 points (maximum impairment). A higher score indicates a worse outcome. Population: Baseline characteristics data from the external placebo arm of the APOLLO study was not summarized with the data from HELIOS-A. APOLLO placebo data was only used as an external comparator for the primary and most other efficacy endpoints. Therefore APOLLO placebo baseline characteristic data is reported separately.
  score on a scale
    number analyzed (Participants) | 77 | 0 | 0 | 77
    (all) | 74.61 (37.041) |  |  | 74.61 (37.041)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Modified Neurologic Impairment Score +7 (mNIS+7) at Month 9 Between the Vutrisiran Group (HELIOS-A) and the External Placebo Comparator Group [APOLLO (NCT01960348)]
Description: The mNIS+7 is a composite score that measures neurologic impairment which includes the following components: physical exam of lower limbs, upper limbs and cranial nerves to assess motor strength/weakness, electrophysiologic measurement of small and large nerve fiber function, sensory testing and postural blood pressure. The mNIS+7 is scored from 0 (no impairment) to 304 points (maximum impairment). A higher score indicates a worse outcome.
Time Frame: Baseline, Month 9
Population: Modified Intent-to-Treat (mITT) Population: All randomized participants who received any amount of study drug. Participants were analyzed according to the treatment to which they were randomized.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Vutrisiran + Vutrisiran (HELIOS-A): Participants will receive vutrisiran 25 mg subcutaneous (SC) injection once every 3 months (q3M) for 18 months during the Treatment Period followed by vutrisiran SC injection during the Randomized Treatment Extension (RTE) Period.
Arm/Group | External Placebo Comparator (APOLLO) | Vutrisiran + Vutrisiran (HELIOS-A)
Number analyzed (Participants) | 77 | 122
score on a scale | 14.76 (2.00) | -2.24 (1.43)
Statistical Analysis 1: Comparison: External Placebo Comparator (APOLLO) vs Vutrisiran + Vutrisiran (HELIOS-A); Multiple imputation estimates and p-value derived per combining least squares (LS) estimates per Rubin's rules based on 100 datasets where missing Month 9 values were imputed using a regression procedure including select baseline variables. LS estimates derived from analysis of covariance model, controlling for categorical factors (treatment, genotype, age of disease onset) and continuous covariate (baseline value); Test type: Equivalence — H0: No difference between vutrisiran and external placebo comparator (APOLLO): difference (vutrisiran - placebo) = 0; p < 0.0000001, ANCOVA with Multiple Imputation — P=3.542E-12; LS Mean Difference = -17.00, 95% CI 2-sided [-21.78 to -12.22], Standard Error of Mean 2.44

2. Secondary Outcome: Change From Baseline in Norfolk Quality of Life-Diabetic Neuropathy (Norfolk QoL-DN) Total Score at Month 9 Between the Vutrisiran Group (HELIOS-A) and the External Placebo Comparator Group [APOLLO (NCT01960348)]
Description: The Norfolk QoL-DN questionnaire is a standardized 35-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy - small fiber, large fiber, and autonomic nerve function. The total score ranges from -4 (best possible quality of life) to 136 points (worst possible quality of life). A higher score indicates a worse outcome.
Time Frame: Baseline, Month 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | External Placebo Comparator (APOLLO) | Vutrisiran + Vutrisiran (HELIOS-A)
Number analyzed (Participants) | 77 | 122
score on a scale | 12.9 (2.2) | -3.3 (1.7)
Statistical Analysis 1: Comparison: External Placebo Comparator (APOLLO) vs Vutrisiran + Vutrisiran (HELIOS-A); Multiple imputation estimates and p-value derived per combining least squares (LS) estimates per Rubin's rules based on 100 datasets where missing Month 9 values were imputed using a regression procedure including select baseline variables. LS estimates derived from analysis of covariance model, controlling for categorical factors (treatment, genotype, age of disease onset baseline NIS) and continuous covariate (baseline value); Test type: Equivalence — H0: No difference between vutrisiran and external placebo comparator (APOLLO): difference (vutrisiran - placebo) = 0; p < 0.0000001, ANCOVA with Multiple Imputation — P=5.426E-09; LS Mean Difference = -16.2, 95% CI 2-sided [-21.7 to -10.8], Standard Error of Mean 2.8

3. Secondary Outcome: Change From Baseline in the Timed 10-Meter Walk Test (10-MWT) at Month 9 Between the Vutrisiran Group (HELIOS-A) and the External Placebo Comparator Group [APOLLO (NCT01960348)]
Description: The 10-MWT is a measure of ambulatory ability and measures the time (in seconds) that it takes a participant to walk 10 meters (gait speed). An increase in gait speed from baseline represents improvement, and a decrease from baseline represents worsening.
Time Frame: Baseline, Month 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: m/sec
Arm/Group | External Placebo Comparator (APOLLO) | Vutrisiran + Vutrisiran (HELIOS-A)
Number analyzed (Participants) | 77 | 122
m/sec | -0.133 (0.025) | -0.001 (0.019)
Statistical Analysis 1: Comparison: External Placebo Comparator (APOLLO) vs Vutrisiran + Vutrisiran (HELIOS-A); Multiple imputation estimates and p-value derived per combining least squares (LS) estimates per Rubin's rules based on 100 datasets where missing Month 9 values were imputed using a regression procedure including select baseline variables. LS estimates derived from analysis of covariance model, controlling for categorical factors (treatment, genotype, age of disease onset, baseline NIS) and continuous covariate (baseline value); Test type: Equivalence — H0: No difference between vutrisiran and external placebo comparator (APOLLO): difference (vutrisiran - placebo) = 0; p < 0.0000001, ANCOVA with Multiple Imputation — P=3.103E-05; LS Mean Difference = 0.131, 95% CI 2-sided [0.070 to 0.193], Standard Error of Mean 0.031

4. Secondary Outcome: Change From Baseline in the Modified Neurologic Impairment Score +7 (mNIS+7) at Month 18 Between the Vutrisiran Group (HELIOS-A) and the External Placebo Comparator Group [APOLLO (NCT01960348)]
Description: The mNIS+7 is a composite score that quantifies motor, sensory, and autonomic neurologic impairment due to injury of large and small nerves. The mNIS+7 is scored from 0 (no impairment) to 304 points (maximum impairment). A higher score indicates a worse outcome.
Time Frame: Baseline, Month 18
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Norfolk QoL-DN Total Score at Month 18 Between the Vutrisiran Group (HELIOS-A) and the External Placebo Comparator Group [APOLLO (NCT01960348)]
Description: as for outcome 2
Time Frame: Baseline, Month 18
Reporting Status: Not Posted

6. Secondary Outcome: Change From Baseline in the 10-MWT at Month 18 Between the Vutrisiran Group (HELIOS-A) and the External Placebo Comparator Group [APOLLO (NCT01960348)]
Description: as for outcome 3
Time Frame: Baseline, Month 18
Reporting Status: Not Posted

7. Secondary Outcome: Change From Baseline in the Modified Body Mass Index (mBMI) at Month 18 Between the Vutrisiran Group (HELIOS-A) and the External Placebo Comparator Group [APOLLO (NCT01960348)]
Description: The mBMI, which is a measure of nutritional status, is calculated as the product of body mass index (BMI) (weight in kilograms divided by the square of height in meters) and serum albumin (g/L) to reflect fluid balance, such as fluid accumulation or dehydration. A negative change from baseline indicates a better outcome.
Time Frame: Baseline, Month 18
Reporting Status: Not Posted

8. Secondary Outcome: Change From Baseline in the Rasch-Built Overall Disability Scale (R-ODS) at Month 18 Between the Vutrisiran Group (HELIOS-A) and the External Placebo Comparator Group [APOLLO (NCT01960348)]
Description: The R-ODS is a patient-reported measure of level of disability on a scale of 0-48, with 0 being the worst and 48 the best (no limitations); scores are based on activities of daily living and social participation. An increase in R-ODS from baseline suggests improvement in disability, and a decrease from baseline suggests worsening of disability.
Time Frame: Baseline, Month 18
Reporting Status: Not Posted

9. Secondary Outcome: Percent Reduction in Serum Transthyretin (TTR) Levels Through Month 18 Between the Vutrisiran Group (HELIOS-A) and the Patisiran Group (HELIOS-A)
Description: Serum TTR was assessed at multiple timepoints up to Month 18.
Time Frame: Up to Month 18
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Non-serious AEs from first dose of study drug through Month 9. SAEs from signing of informed consent through Month 9.
Description: Adverse events are provided for the vutrisiran group and the reference comparator (patisiran) group as of the data cutoff date (10 November 2020).
Arm/Group | Vutrisiran + Vutrisiran (HELIOS-A) | Patisiran + Vutrisiran (HELIOS-A)
All-Cause Mortality (participants affected / at risk) | 2/122 | 3/42
Serious Adverse Events (participants affected / at risk) | 21/122 | 17/42
Other Adverse Events (participants affected / at risk) | 78/122 | 31/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vutrisiran + Vutrisiran (HELIOS-A) (N=122) | Patisiran + Vutrisiran (HELIOS-A) (N=42)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Infusion site phlebitis (General disorders) | 0 | 1
Infusion related reaction (Immune system disorders) | 0 | 3
COVID-19 (Infections and infestations) | 2 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 1
Endocarditis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Infusion site cellulitis (Infections and infestations) | 0 | 2
Kidney infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Cardiovascular evaluation (Investigations) | 0 | 1
Investigation (Investigations) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Endometrial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Iliac artery occlusion (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vutrisiran + Vutrisiran (HELIOS-A) (N=122) | Patisiran + Vutrisiran (HELIOS-A) (N=42)
Abdominal pain (Gastrointestinal disorders) | 7 | 0
Constipation (Gastrointestinal disorders) | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 15 | 4
Nausea (Gastrointestinal disorders) | 11 | 4
Vomiting (Gastrointestinal disorders) | 7 | 3
Oedema peripheral (General disorders) | 10 | 4
Infusion related reaction (Immune system disorders) | 0 | 9
Nasopharyngitis (Infections and infestations) | 8 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 4
Urinary tract infection (Infections and infestations) | 13 | 5
Fall (Injury, poisoning and procedural complications) | 12 | 4
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 3
Alanine aminotransferase increased (Investigations) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 3
Vitamin A decreased (Investigations) | 8 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 4
Dizziness (Nervous system disorders) | 9 | 0
Headache (Nervous system disorders) | 8 | 5
Neuralgia (Nervous system disorders) | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is intended that after completion of the study, the data are to be submitted for publication in a scientific journal and/or for reporting at a scientific meeting. A copy of any proposed publication (eg, manuscript, abstracts, oral/slide presentations, book chapters) based on this study, must be provided and confirmed/received at the Sponsor at least 30 days before its submission.

DOCUMENTS (2):
  • Study Protocol (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT03759379/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT03759379/SAP_001.pdf